CLINICAL TRIAL: NCT03498976
Title: Evaluation of Pulsed Radiofrequency on the Suprascapular Nerve Versus Radiofrequency Pulsed on Suprascapular Nerve and Circumflex in the Treatment of Painful Shoulder
Brief Title: RFp on Suprascapular N. Versus RFp on Suprascapular N. and Circumflex in the Treatment of Painful Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP-RF
Record Dates: First submitted 2018-03-28; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Pain Syndrome
Keywords: painful shoulder
MeSH Terms: conditions — Somatoform Disorders | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed radiofrequency on SE nerve (Other): Single technic
  Interventions: Procedure: pulsed radiofrequency
- Pulsed radiofrequency on SE + CF nerves (Other): Combinated technic
  Interventions: Procedure: pulsed radiofrequency

INTERVENTIONS:
Procedure: pulsed radiofrequency — Echoguided technic

SUMMARY:
Pulsed radiofrequency produces more lasting pain relief than use of peripheral blocks or analgesic medication in the treatment of chronic pain.

We study the use of pulsed radiofrequency on the suprascapular nerve and the Circumflex nerve and the efficacy of the single technique on suprascapular nerve versus the circumflex and suprascapular combinated technique

DETAILED DESCRIPTION:
The painful shoulder is responsible for approximately 16% of all musculoskeletal complaints, constituting one of the most frequent consultations in primary care only behind patients with low back and neck pain.

It has been estimated that 20% of the general population will suffer shoulder pain throughout their lives with a prevalence that can reach up to 50%. It is more prevalent in the elderly with 21% and up to 20% in diabetic patients.

The "painful shoulder syndrome" is a frequent and disabling pathology, of diverse etiology and complex diagnosis, being more common in the female population, and especially from the fifth decade of life in an age range between 45-65 years, although it may manifest itself in other age groups. The prevalence increases with age, some professions and certain sports activities.

Between 70% and 85% of consultations are due to rotator cuff pathology, the most frequent cause of shoulder pain being inflammation of the tendons that form it (supraspinatus, subscapularis, infraspinatus, teres minor and the long portion of the biceps). These are extra-articular muscles, so the clinical picture is called scapulohumeral periarthritis.

Objectives:

Main objective To evaluate the degree of decrease in pain assessment scales (VAS) and decrease in disability scale (SPADI).

Secondary objectives I. Measure the time during which the patient improves pain. II. Evaluate the improvement in the Constant Murley range of motion scale. III. Analyze the recovery in the functionality of the shoulder and performing basic activities of daily living (DASH scale).

IV. Analyze the decrease in the need for analgesic medication (NSAIDs and opiates).

V. Assess the appearance of complications related to the performance of pulsed radiofrequency guided with ultrasound.

Study design The patients were evaluated following the usual protocol of the Pain Unit in which all demographic data, age, sex, reason for consultation, personal history, history of pain, exploration and proposed treatment as well as the complementary tests performed were collected. With the clinical judgment of painful shoulder syndrome, if it met at least one inclusion criterion (table), the patient was exposed to the therapeutic possibilities and the possibility of entering the study.

Subsequently, in a period of no more than 30 days, the interventionist technique is performed in the Pain Unit technique room. Finally, a clinical follow-up is carried out in consultation with the Pain Unit at month, three months, six months and nine months from the date of completion of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Frozen shoulder syndrome (adhesive capsulitis) of more than 3 months evolution Massive rotator cuff tear Partial rupture of some tendon of the rotator cuff Arthrosis of the joint Humeral scapular periarthritis Calcifying tendinitis Bursitis Subacromial syndrome operated by shoulder arthroscopy and persistence of pain over 3 months evolution

Exclusion Criteria:

* Rejection of the realization of the technique Anticoagulation or active coagulopathies Infection at the puncture site Psychopathologies or psychiatric problems Judicial litigation at the beginning of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-25 (Estimated)

PRIMARY OUTCOMES:
Degree of decrease in pain assessment scales (VAS) | 9 MONTHS
  Change From Baseline on the VAS

SECONDARY OUTCOMES:
Degree of SPADI scale improvement | 9 MONTHS
  Change From Baseline in SPADI scale
Improvement in the Constant Murley range of motion scale. | 9 MONTHS
  Change From Baseline in Constant Murley range of motion scale
Recovery in the functionality of the shoulder and performing basic activities of daily living (DASH scale). | 9 MONTHS
  Change From Baseline in DASH scale

CONTACTS AND LOCATIONS:
Overall Officials: JOSÉ MIGUEL ESPARZA MIÑANA, MD, Principal Investigator — Hospital de Manises
Locations (1):
- José Miguel Esparza Miñana, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
WORK IN PROCESS